CLINICAL TRIAL: NCT03102294
Title: Inspiratory Muscle Training in Patients With Pulmonary Hypertension: a Double-blind Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Roberta Pulcheri Ramos, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUSaoPaulo2017
Record Dates: First submitted 2017-03-22; First posted 2017-04-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Inspiratory Muscle Training; Inspiratory Muscle Weakness; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: IMT (Active Comparator): inspiratory muscle training (PowerBREATHE) with ~50% of maximum inspiratory pressure
  Interventions: Other: inspiratory muscle training
- Placebo: SHAM (Placebo Comparator): inspiratory muscle training (PowerBREATHE) without inspiratory load
  Interventions: Other: Placebo "training"

INTERVENTIONS:
Other: inspiratory muscle training — inspiratory muscle training with 50% of MIP
  Arms: Experimental: IMT
Other: Placebo "training" — placebo training with PowerBreathe (without inspiratory load)
  Arms: Placebo: SHAM

SUMMARY:
Inspiratory muscle training for 8 weeks in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
32 patients with PH will perform: 1) pulmonary function tests; 2) measurement of maximal inspiratory pressure (MIP) and endurance; 3) six-minute walk test and 5) incremental and constant load cardiopulmonary exercise test (~ 75% of maximal work-rate) and step test. Inspiratory muscle training will consist of twice daily sessions of 30 breaths (~ 50% PiMAX, 4-5 minutes per session) for 8 weeks. The SHAM group will perform sessions of 30 breaths with no inspiratory load.

ELIGIBILITY:
Inclusion Criteria:

* CTEPH confirmed by RHC and imaging
* NYHA FC II-IV

Exclusion Criteria:

* Limitation to cycling
* Recent syncope or clinical deterioration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
exercise capacity¨- cardiopulmonary exercise testing | week 8
  TLim (seconds)
exercise capacity - 6-min walk test | week 8
  distance (m)

SECONDARY OUTCOMES:
ventilatory responses | Week 8
  VE/VCO2

CONTACTS AND LOCATIONS:
Locations (1):
- SEFICE - Setor de Função Pulmonar e Fisiologia Clínica do Exercício, São Paulo, São Paul, Brazil

IPD SHARING:
Plan to Share IPD: Yes